CLINICAL TRIAL: NCT03522948
Title: Alcohol and Implicit Process in Sexual Risk Behavior in MSM- Supplement
Brief Title: Alcohol and Sex Risk Intervention for MSM Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Tibor Palfai, Professor of Psychological and Brain Sciences, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3468; 3R01AA022301-02S1 (NIH)
Record Dates: First submitted 2018-04-18; First posted 2018-05-14 (Actual); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Heavy Drinking and Sexual Risk Behavior
Keywords: heavy drinking; sexual risk behavior
MeSH Terms: interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Open pilot study to test feasibility of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open pilot (Experimental): The intervention is a brief, in-person motivational intervention followed by 4 weeks of text messaging to reduce heavy episodic drinking and sexual risk behavior (unprotected anal intercourse) among men-who-have-sex-with-men.
  Interventions: Behavioral: Brief intervention with text messaging to reduce sexual risk and heavy drinking among MSM

INTERVENTIONS:
Behavioral: Brief intervention with text messaging to reduce sexual risk and heavy drinking among MSM — Combines a brief in-person motivational intervention with personalized cognitive counseling elements and 4 weeks of personalized text messaging to support goals related to sexual risk behavior and alcohol use
  Other Names: Intervention to reduce heavy drinking and sex risk among MSM

SUMMARY:
Open pilot trial to test the feasibility and efficacy of a brief intervention with text messaging to reduce sexual risk behavior and heavy drinking among MSM

DETAILED DESCRIPTION:
This study seeks to develop and provide an initial test of a brief intervention to reduce alcohol use and sex risk behavior among among men who have sex with men. The study seeks to recruit MSM who are non-monogamous, have engaged in unprotected anal intercourse over the past 3 months, and who have engaged in heavy drinking defined as > 14 drinks per week or at least 1 heavy drinking episode (5+ drinks on a single occasion) in the past month. All participants will complete baseline measures about past month behavior and if eligible will be assigned to the intervention condition. This intervention consists of a single brief in-person intervention coupled with 4 weeks of text messaging related to individualized goals about alcohol use and sexual behavior. Follow-up assessments are scheduled for within 1 week of completion of the text messaging component of the intervention. Primary outcomes are feasibility and acceptability of the intervention and message components. Secondary outcomes are changes in frequency of unprotected intercourse and heavy drinking episodes.

ELIGIBILITY:
Inclusion Criteria:

Non-monogamous bisexual/gay male with Kinsey score indicating mainly homosexual identification, heavy drinking, UAI in past 3 months.

-

Exclusion Criteria:

HIV+ Past or current tx for alcohol use (past 3 years), bipolar disorder or schizophrenia Current psychiatric treatment Medications contraindicated by alcohol Medical conditions contraindicated by alcohol Substance specific ASSIST scores of 27 or greater

-

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Palfai, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Pilot
Started | 8
Completed | 7
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Pilot
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (2.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Intervention Satisfaction Scale
Description: 3-item modification of Client Satisfaction Questionnaire. Three 5-point Likert scale is used to assess "intervention satisfaction" [very dissatisfied - very satisfied]; degree to which intervention helped alcohol use [no effect to helped a great deal], and intervention helped sexual behavior decisions [no effect - helped a great deal]. Mean scale range is 1-5. Higher scores reflect a better outcome
Time Frame: Participants complete the measure 5-6 weeks following baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Pilot
Number analyzed (Participants) | 7
units on a scale | 4.25 (0.05)

2. Secondary Outcome: Frequency of Heavy Episodic Drinking Measure From the Alcohol Use Disorders Identification Test
Description: This measure is a 5-point Likert scale item which asks participants to report "How often do you have six or more drinks on one occasion?" Response options range from "never" to "daily or almost daily." This measure is completed at baseline and 5 to 6 weeks after baseline. Higher scores reflect worse outcomes. Responses reflect current perceptions of past drinking. Range 0-4
Time Frame: Participants report frequency of heavy drinking episodes as part of the AUDIT-C questionnaire. The question is presented at baseline and at follow-up which occurs 5-6 weeks following baseline. There is no timeframe specified in the question itself.
Population: computer processing error lead to omission of 2 participants for this analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Pilot
Number analyzed (Participants) | 5
score on a scale
  Baseline | 2.60 (0.55)
  Follow-up | 1.60 (0.55)
Statistical Analysis 1: Comparison: Open Pilot; within-subject t-test; Test type: Superiority; p = .03, t-test, 2 sided; Mean Difference (Net) = -3.16, Standard Deviation -.71

3. Secondary Outcome: Frequency of Condomless Anal Intercourse.
Description: Single item measure of number of times that individual engaged in unprotected intercourse. Range is 0-30 for baseline (reflecting 0-90 range for past 3 months divided by 3) and range is 0-30 for follow-up. Higher scores reflect a worse outcome.
Time Frame: Frequency of condomless anal intercourse (CAI) over the past 3 months at baseline (divided by 3 for monthly CAI) and rate frequency of condomless anal intercourse over the past month at follow-up assessment that occurs 5-6 weeks following baseline.
Measure: Mean (Standard Deviation); unit: condomless anal intercourse
Arm/Group | Open Pilot
Number analyzed (Participants) | 7
condomless anal intercourse
  Baseline Monthly CAI | 2.67 (1.35)
  Follow-Up past Month CAI | 1.29 (1.38)
Statistical Analysis 1: Comparison: Open Pilot; Test type: Superiority; p = 0.23, t-test, 2 sided; t-test = -1.34, Standard Deviation 3.20; d = -0.51

4. Post Hoc Outcome: Goal Systems Assessment Battery (Karoly & Ruehlman, 1995) for Behavior Goal of "Reducing Alcohol Use".
Description: This GSAB battery consists of 4 subscales comprised of 4 Likert-scale items each ranging from 0-4. The subscales indicate value, self-efficacy, monitoring and planning related to the behavior change goal of reducing alcohol use. The mean subscale range is from 0-16. Higher scores reflect better self-regulatory outcomes.
Time Frame: This measure was taken at baseline and at follow-up. There is no specific timeframe indicated in the measure as it is used to indicate current goal cognitions. The measure is completed at baseline and 5 to 6 weeks following baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Pilot
Number analyzed (Participants) | 7
units on a scale
  Baseline GSAB Reducing Alcohol -Value | 5.71 (2.69)
  Follow-up GSAB Reducing Alcohol Value | 10 (3.61)
  Baseline GSAB Reducing Alcohol Self-Efficacy | 12.14 (2.48)
  Follow-up GSAB Reducing Alcohol Self-Efficacy | 13 (2.71)
  Baseline GSAB Reducing Alcohol Self-Monitoring | 6.14 (4.14)
  Follow-up GSAB Reducing Alcohol Self-Monitoring | 9.71 (2.63)
  Baseline GSAB Reducing Alcohol Planning | 4.86 (4.26)
  Follow-up GSAB Reducing Alcohol Planning | 8.14 (3.24)
Statistical Analysis 1: Comparison: Open Pilot; GSAB self-efficacy; Test type: Superiority; p < .05, t-test, 2 sided; t-test = 1.35, 95% CI 2-sided [-0.69 to 2.41]

5. Post Hoc Outcome: Goal Systems Assessment Battery (Karoly & Ruehlman, 1995) for Behavior Goal of "Using Condoms Every Time You Have Sex With a Partner of Unknown HIV Status".
Description: This GSAB battery consists of 4 subscales comprised of 4 Likert scale items each ranging from 0-4. Items are summed to create subscale scores. The subscales indicate value, self-efficacy, planning, and monitoring related to the behavior change goal. The mean subscale range is from 0-16. Higher scores reflect better self-regulatory outcomes
Time Frame: This measure was taken at baseline and at follow-up. There is no specific timeframe indicated on the questions as the measure indicates current goal cognitions. The measure is completed at baseline and 5 to 6 weeks following baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Pilot
Number analyzed (Participants) | 7
units on a scale
  Baseline GSAB Condom Value | 11.14 (5.52)
  Follow-up GSAB Condom Value | 13.71 (2.21)
  Baseline GSAB Condom Self-Efficacy | 11.57 (3.36)
  Follow-up GSAB Condom Self-Efficacy | 13.43 (2.70)
  Baseline GSAB Condom Self-Monitoring | 7.29 (4.96)
  Follow-up GSAB Condom Self-Monitoring | 11.14 (3.85)
  Baseline GSAB Condom Planning | 7.43 (5.38)
  Follow-up GSAB Condom Planning | 11.43 (3.64)
Statistical Analysis 1: Comparison: Open Pilot; Test of GSAB self-efficacy subscale for condom use; Test type: Superiority; p < .05, t-test, 2 sided; t-test = 2.93, 95% CI 2-sided [0.31 to 3.41]

ADVERSE EVENTS:
Time Frame: through study completion, up to six weeks
Arm/Group | Open Pilot
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
The focus of the intervention was feasibility and acceptability, not results of inferential statistical analysis as this is a small sample in an open pilot

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT03522948/Prot_SAP_000.pdf